CLINICAL TRIAL: NCT05949281
Title: Repurposing Colchicine for Reduction of Residual Inflammatory Risk in Type 1 Diabetes: A Randomized, Double-blind, Placebo-controlled, Investigator-initiated Trial
Brief Title: Repurposing Colchicine for Reduction of Residual Inflammatory Risk in Type 1 Diabetes
Acronym: REC1TE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asger Lund, MD (Other)
Collaborators: University of Copenhagen (Other); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Asger Lund, MD, Ass. Professor, MD, PhD, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-502038-23-00
Record Dates: First submitted 2023-06-29; First posted 2023-07-18 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes; Cardiovascular Diseases; Chronic Inflammation
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Cardiovascular Diseases | interventions — Colchicine; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Active Comparator): Colchicine tablet 0.5 mg once-daily
  Interventions: Drug: Colchicine 0.5 MG Oral Tablet
- Placebo (Placebo Comparator): Placebo tablet once-daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Colchicine 0.5 MG Oral Tablet — Colchicine 0.5 mg once-daily
  Other Names: Colrefuz
  Arms: Colchicine
Drug: Placebo — Placebo tablet once-daily
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to evaluate if colchicine in addition to standard of care improves markers of inflammation and cardiovascular disease in persons with type 1 diabetes. Participants will be assigned to either 0,5 mg colchicine daily or placebo in a 1:1 ratio for 26 weeks with the possibility of an additional 26 week extension of the intervention period. After the treatment period, there will a 5-year follow-up on all available outcome measures via electronic patient records for those who took part in the extension.

DETAILED DESCRIPTION:
The current study aims to evaluate the efficacy of 0.5 mg colchicine once-daily added to existing standard of care in persons with established type 1 diabetes, existing arteriosclerotic cardiovascular disease (CVD) or at high risk thereof and C-reactive protein (CRP) ≥ 2 mg/L. Specifically, the primary objective is to determine the effect of colchicine (0.5 mg/daily) on levels of CRP (as assessed by high-sensitivity assays) as compared with placebo following 26-52 weeks of treatment. Additionally, the study will investigate the short and long-term effects of colchicine treatment on other markers of CVD and inflammation, markers of metabolism and markers of glycemic control in type 1 diabetes, including glycated hemoglobin (HbA1c), time spent in hypoglycemia (level 1 glucose readings 3.0-3.8 mmol/L and level 2 glucose readings < 3.0 mmol/L), target glycemia (glucose readings 3.9-10 mmol/L) and hyperglycemia (level 1 glucose readings 10.1-13.9 mmol/L and level 2 glucose readings > 13.9 mmol/L) together with measures of glycemic variability evaluated by continuous glucose monitoring (CGM), insulin dosage, risk of hypoglycemia, risk of diabetic ketoacidosis and body weight. During the 5-year follow-up, we will collect all available outcome measures via electronic patient records.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for more than five years according to World Health Organization criteria
* Age 35-80 years
* Hemoglobin A1c < 80 mmol/mol
* Stable insulin therapy (defined as no change in insulin brand and no newly initiated continous subcutaneus insulin infusion (CSII) or multiple-daily injection (MDI) therapy) and, if applicable, stable usage of glucose monitoring technology (e.g., continous glucose monitor (CGM) or intermittently scanned CGM) ≥ 3 months with either MDI or CSII
* CRP ≥ 2 mg/L (measured by high-sensitivity assay)
* eGFR > 50 mL/min/L/1.73 m^2
* Either stable arteriosclerotic cardiovascular disease (ASCVD) (as defined by ischemic heart disease including previous acute myocardial infarction, acute coronary syndrome and coronary revascularization; other arterial revascularization procedures; stroke and transient ischemic attack; aortic aneurysm; peripheral arterial disease, including carotid atherosclerosis)
* and/or risk of cardiovascular (CV) death > 5 % within 10 years (i.e., high or very high CV risk) as defined by the European Society of Cardiology or 10-year CV risk ≥ 20 % (i.e., high CV risk) as according to 'Steno Type 1 Diabetes Risk Engine' (https://steno.shinyapps.io/T1RiskEngine/)

Exclusion Criteria:

* Hypoglycemia unawareness (inability to register low blood glucose) am modum Pedersen-Bjergaard, unless usage of CGM with alarm function
* Liver disease with elevated plasma alanine aminotransferase (ALT) > three times the upper limit of normal (measured at screening with the possibility of one repeat analysis within seven days, and the last measured value as being conclusive)
* History of cirrhosis, chronic active hepatitis or severe hepatic disease
* Inflammatory bowel disease or chronic diarrhea
* Pre-existing progressive neuromuscular disease or persons with creatinine kinase levels > three times the upper limit of normal (measured at screening with the possibility of one repeat analysis within a week, and the last measured value as being conclusive)
* Cancer or lymphoproliferative disease unless in complete remission for > 5 years
* Immunosuppressive therapy or state of chronic immunodeficiency, including infection with human immunodeficiency virus (HIV)
* Blood dyscrasias (e.g., myelodysplastic syndromes or related hematological disorders)
* Leukocyte cell count < 3.0 X 10^9/L
* Thrombocyte count < 110 X 10^9/L
* Systemic (oral or intravenous), long-term steroid therapy (topical or inhaled steroids are allowed)
* Hemodialysis or peritoneal dialysis therapy (since colchicine cannot be removed by dialysis or exchange transfusion)
* Renal or hepatic impairment treated with a P-gp inhibitor or a strong CYP3A4 inhibitor
* Intake of grapefruit juice during trial participation
* Other concomitant disease or treatment that according to the investigator's assessment makes the person unsuitable for study participation
* Alcohol/drug abuse
* Fertile women not using hormonal (tablet/pill, depot injection of progesterone, subdermal gestagen implantation, hormone intrauterine devices (IUD), hormonal vaginal ring or transdermal hormonal patch), chemical (copper IUD) or mechanical (condom, femidom, sterilization) contraceptives
* Pregnant or nursing women
* On permanent treatment with colchicine that is not discontinued within 30 days of screening visit
* Known or suspected hypersensitivity to colchicine
* Receipt of any investigational drug within 30 days prior to screening visit
* Simultaneous participation in any other clinical intervention trial

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2031-01-15 (Estimated); Study Completion 2031-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in fasting serum/plasma concentrations of C-reactive protein (CRP) measured by a high-sensitivity assay (hsCRP) (mg/L) | From week 0 (baseline) to week 26 (end of treatment)
  %-point

SECONDARY OUTCOMES:
Change in fasting serum/plasma concentrations of C-reactive protein (CRP) measured by a high-sensitivity assay (hsCRP) (mg/L) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of hemoglobin A1c (mmol/mol) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Time spent in target blood glucose range (3.9 - 10 mmol/L) evaluated by a continous glucose monitor (CGM) | From week 0 (baseline) to week 26 (end of treatment) or to 52 weeks (extension)
  (% of 24 hours)
Time spent in hyperglycemia level 1 (10-13.9 mmol/L) evaluated by a continous glucose monitor (CGM) | From week 0 (baseline) to week 26 (end of treatment) or to 52 weeks (extension)
  (% of 24 hours)
Time spent in hyperglycemia level 2 (> 13.9 mmol/L) evaluated by a continous glucose monitor (CGM) | From week 0 (baseline) to week 26 (end of treatment) or to 52 weeks (extension)
  (% of 24 hours)
Time spent in hypoglycemia level 1 (3.0-3.8 mmol/L) evaluated by a continous glucose monitor (CGM) | From week 0 (baseline) to week 26 (end of treatment) or to 52 weeks (extension)
  (% of 24 hours)
Time spent in hypoglycemia level 2 (< 3.0 mmol/L)evaluated by a continous glucose monitor (CGM) | From week 0 (baseline) to week 26 (end of treatment) or to 52 weeks (extension)
  (% of 24 hours)
Insulin dosage | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  Number of units/day (both long- and short-acting insulin analogues)
Change in body weight (kg) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in waist:hip ratio | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of low-density lipoprotein cholesterol (LDL) (mmol/L) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of interleukin (IL)-6 (pg/mL) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of tumor necrosis factor alpha (pg/mL) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Safety-related events | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  Serious adverse events (SAE), events of severe hypoglycemia, events of diabetic ketoacidosis

OTHER OUTCOMES:
Change in fasting serum/plasma concentrations of fibrinogen (µmol/L) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of serum amyloid A (mg/L) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of haptoglobin (g/L) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of interleukin (IL)-1β (pg/mL) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of interleukin (IL)-2 (pg/mL) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of intercellular adhesion molecule 1 (ICAM-1) (pg/mL) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of vascular cell adhesion molecule 1 (VCAM-1) (pg/mL) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of total leukocyte count, including neutrophil, lymphocyte, basophil and eosinophil counts (10^9/L) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in neutrophil:lymphocyte ratio | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of very low-density lipoprotein (VLDL) cholesterol (mmol/L) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of high-density lipoprotein (HDL) cholesterol (mmol/L) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of total cholesterol (mmol/L) | From week 0 (baseline) to week 30 (safety follow-up) or to 56 weeks (extension)
  %-point
Change in fasting serum/plasma concentrations of triglycerides (mmol/L) | From week 0 (baseline) to week 30 (safety follow-up) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of lipoprotein (a) (mg/L) | From week 0 (baseline) to week 30 (safety follow-up) or to week 56 (extension)
  %-point
Change in thrombocyte function measured by thromboelastography | From week 0 (baseline) to week 26 (end of treatment) or to week 52 (extension)
  %-point
Change in fasting serum/plasma concentrations of N-terminal pro-brain natriuretic peptide (pro-BNP) (pmol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in consultation blood pressure (mmHg) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in heart rate (beats/minute) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of estimated glomerular filtration rate (eGFR) (mL/min/1.73 m2) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of albumin (g/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in urine albumin-to-creatinine ratio (mg/g) | From week 0 (baseline) to week 26 (end of treatment) or to week 56 (extension)
  %-point
Change left ventricular (LV) mass index evaluated by cardiovascular ultrasonography (g/m^2) | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change left ventricular (LV) septal wall thickness evaluated by cardiovascular ultrasonography (mm) | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change left ventricular (LV) posterior wall thickness evaluated by cardiovascular ultrasonography (mm) | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change left ventricular (LV) ejection fraction (LVEF) evaluated by cardiovascular ultrasonography (%) | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change ratio of peak velocity blood flow from left ventricular relaxation in early diastole (E) to peak velocity flow in late diastole caused by atrial contraction (A) (E/A ratio) evaluated by cardiovascular ultrasonography | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change early diastolic mitral inflow velocity (e') evaluated by cardiovascular ultrasonography (m/sec) | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change ratio of early diastolic mitral inflow velocity (e') to early diastolic mitral annulus velocity (E) (E/e' ratio) evaluated by cardiovascular ultrasonography | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change ratio of early mitral inflow velocity (E) to global diastolic strain rate (e' sr) (E/e'sr ratio) evaluated by cardiovascular ultrasonography | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change left atrial volume (LAVi) evaluated by cardiovascular ultrasonography (mL) | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change global longitudinal strain (GLS) evaluated by cardiovascular ultrasonography (%) | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change aortic distensibility evaluated by cardiovascular ultrasonography (mmHg^-1) | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change aortic strain evaluated by cardiovascular ultrasonography (%) | From week 0 (baseline) to week 26 (end of treatment)
  %-point
Change in mean glucose evaluated by a continous glucose monitor (mmol/L) | From week 0 (baseline) to week 26 (end of treatment) or to week 52 (extension)
  %-point
Change in standard deviation evaluated by a continous glucose monitor (mmol/L) | From week 0 (baseline) to week 26 (end of treatment) or to week 52 (extension)
  %-point
Change in coefficient of variance evaluated by a continous glucose monitor (> 0.36 defined as glycemic variability) | From week 0 (baseline) to week 26 (end of treatment) or to week 52 (extension)
  %-point
Change in glycemic variability (continuous overall net glycemic action (CONGA)) evaluated by a continous glucose monitor | From week 0 (baseline) to week 26 (end of treatment) or to week 52 (extension)
  %-point
Change in mean amplitude of glycemic excursion evaluated by a continous glucose monitor | From week 0 (baseline) to week 26 (end of treatment) or to week 52 (extension)
  %-point
Change in diabetes treatment satisfactory questionnaire, status version (DTSQs) (From 0 (min) to 6 (max), higher scores indicate a better outcome ) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in diabetes treatment satisfactory questionnaire, change version (DTSQc) (From -3 (min) to 3 (max), higher scores indicate a better outcome) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in audit of diabetes-dependent quality of life questionnaire (ADDQoL) (From -9 (min) to 9 (max), higher scores indicate a better outcome ) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of ketones (mmol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Adverse events | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  As reported by participants
Change in liver fat content as per the CAP score (dB/m) measured by FibroScan® | From week 0 (baseline) to week 26 (end of treatment) or to week 52 (extension)
  %-point
Change in liver fibrosis score (kPa) measured by FibroScan® | From week 0 (baseline) to week 26 (end of treatment) or to week 52 (extension)
  %-point
Change in fibrosis-4 (FIB-4) score (numerical scale, higher scores indicate a higher risk of fibrosis) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fatty liver index (FLI) score (numerical scale, higher scores indicate a higher risk of fibrosis) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of hemoglobin (mmol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of thrombocytes (10^9/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of glucose (mmol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of potassium (mmol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of sodium (mmol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of creatinine (umol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of alanine aminotransferase (U/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of aspartate aminotransferase (U/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of bilirubin (umol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of amylase (units/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of creatine kinase (U/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of C-peptide (pmol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of glucagon (pmol/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of C-terminal telopeptide (ng/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in fasting serum/plasma concentrations of procollagen type 1 N-terminal propeptide (ng/L) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in body composition by bioimpedance analysis | From week 0 (baseline) to week 26 (end of treatment) or to week 52 (extension)
  %-point (fat free mass, total fat mass, muscle mass, bone mass)
Change in body mass index (kg/m^2) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in waist circumference (cm) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in hip circumference (cm) | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in waist:hip ratio | From week 0 (baseline) to week 30 (end of treatment) or to week 56 (extension)
  %-point
Change in interleukin messenger ribonucleic acid (mRNA) expression measured by quantitative polymerase chain reaction | From week 0 (baseline) to week 26 (end of treatment) or to week 56 (extension)
  %-point

CONTACTS AND LOCATIONS:
Overall Officials: Asger B. Lund, MD, PhD, Principal Investigator — Center for Clinical Metabolic Research, Gentofte Hospital, Denmark
Locations (1):
- Center for Clinical Metabolic Research, Gentofte Hospital, Hellerup, Capital Region, Denmark